CLINICAL TRIAL: NCT03664414
Title: Pentoxifylline Effect on Renal Function, Oxidative Stress, Inflammation, and Fibrosis Markers, and Quality of Life in Patients With Diabetic Nephropathy
Brief Title: Pentoxifylline Effect in Patients With Diabetic Nephropathy.(PENFOSIDINE STUDY)
Acronym: PENFOSIDINE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Eugenia Galván Plata (Other Government)
Collaborators: Centro de Investigación Biomédica de Michoacán. (Unknown); Hospital General Regional N° 1 Instituto Mexicano del Seguro Social. (Unknown); Hospital General de Zona N° 83 Instituto Mexicano del Seguro Social. (Unknown); Coordinación Auxiliar Medica de Investigación en Salud. Delegación Michoacán. (Unknown)
Responsible Party: Sponsor-Investigator, Maria Eugenia Galván Plata, Coordinacion de Investigacion en Salud, México, Coordinación de Investigación en Salud, Mexico
Organization: Coordinación de Investigación en Salud, Mexico (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNIC-2015-785-065
Record Dates: First submitted 2018-07-25; First posted 2018-09-10 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Chronic Kidney Disease stage3 and 4; Type 2 Diabetes Mellitus
Keywords: oxidative stress; fibrosis; inflammation; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fibrosis; Inflammation | interventions — Pentoxifylline

STUDY DESIGN:
Intervention Model Description: blinded,multicenter, randomized, pentoxifylline vs placebo controlled clinical trial. Time: two years after the enrollment of the last patient.
Who Masked: Participant, Investigator
Masking Description: Plaebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator): Placebo group will receive 1 tablet of cellulose pill to mimic pentoxifylline tablets three times a day with meals, during the following two years.
  Interventions: Drug: pentoxifylline
- Pentoxifylline group (Active Comparator): Pentoxifillyne or experimental group will receive 400 mg of pentoxifylline three times a day with meals, during the following two years.
  Interventions: Drug: pentoxifylline

INTERVENTIONS:
Drug: pentoxifylline — Pentoxifylline or placebo will be prescribed three times a day with meals. All the participants will continue with the usual treatment. Time frame: two years
  Other Names: Trental

SUMMARY:
One of the purposes of the management of the patient with chronic kidney disease (CKD)is to slow the decline of renal function. The mechanisms by which the renal function declines involve inflammatory and fibrotic responses due in part by the effects of oxidative stress. Pentoxifylline (PTX)is a drug that stimulates adenosine receptors, and produces inhibition of phosphodiesterases, as well as being a dopaminergic modulator through D1 and D2 receptors. Its main effects are inhibition of the inflammatory state by decreasing serum levels of tumor necrosis factor alpha (TNF-ɒ) and monocyte chemo attractant protein 1 (MCP_1), which may slow down the decline of renal function. It also produces diminish of sympathetic activity, with the reduction of circulating levels of norepinephrine (NA), which may contribute to the reduction of glomerulosclerosis in diabetic patients. In the connective tissue increases the activity of the collagenases and decrease of collagen, fibronectin and glucosamine of the fibroblasts as well as inhibition of oxygen free radicals. Due to its antioxidant, anti-inflammatory and anti-fibrotic effects, PTX can result in an excellent therapeutic option for the prevention of CKD in DM2.

This work proposes the use of pentoxifylline as treatment CKD in DM2. Its application in patients with CKD will allow a therapeutic management with different targets, for its antioxidant, anti-inflammatory and antifibrotic effects that will be evaluated by means of fibrosis, inflammation and oxidative stress markers. The results will be of great importance in clinical practice, since they will justify the use of a new pharmacological tool, already known, with minimal adverse effects and low cost, accessible to all strata of the population since it is found as generic.

DETAILED DESCRIPTION:
Patients will be randomly selected from the outpatient family medicine clinics. Once included, patients will be randomly allocated (by a computer-generated randomization list) to a study or control group. Over a period of 2 years, patients of the study group will receive one PTX tablet (400 mg) orally three times a day (at dinner time), whereas controls will receive one cellulose identical tablet on the same schedule.

All patients will continue with their usual treatment prescribed by their family doctor. Monthly visits will be scheduled for clinical and biochemical evaluations. A blood sample will be taken at baseline and every six months up to 24 months, for measurement of complete blood count, urea, creatinine, glucose, albumin, lipids, electrolytes, liver function tests, serum total proteins, (will be measure by usual methods). In serum samples at 0, 6, 12, 18 and 24 months, high sensibility C reactive protein will be measured by nephelometry, Brain natriuretic peptide and Serum Cystatin C will be measured by ELISA. Glomerular filtration rate (GFR) will be calculated based in Cystatin C level Grubb's equations. Vitamin C will be measured by HPLC. A 24 h ambulatory blood pressure monitoring (24 h ABPM), M-mode and two-dimensional echocardiographic, and an analysis of body composition by bioelectrical impedance will be done at baseline 6, 12, 18 and 24 months. To investigate health-related quality of life the short-form 36 (SF-36) questionnaire will be applied. Treatment compliance will be recorded by counting tablets left in the container at the end of each monthly visit and by the Morinsky Green test.

ELIGIBILITY:
Inclusion Criteria:

1. CKD
2. Type 2 diabetes mellitus
3. Microalbuminuria
4. Proteinuria.
5. Creatinine plasma clearance ˂ of 60 mL / min.

Exclusion criteria:

1. History of psychiatric disorders,
2. Immunosuppressants treatment
3. Herbalism Treatment
4. History of chronic alcoholism.
5. Type 1 diabetes mellitus.
6. Chronic obstructive pulmonary disease.
7. Pulmonary fibrosis
8. Heart failure
9. HIV-AIDS.
10. Liver cirrhosis.
11. Chronic hepatitis.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the glomerular filtration rate | The measurements will be done baseline and every six months up to 24 months.
  It will be measure as to duplicate serum creatinine levels from baseline (mg/dL), or to pass from a stage of chronic kidney disease to he next stage (GFR mL/min)

SECONDARY OUTCOMES:
Change in oxidative stress marker. | Change is assessed baseline, 6 months, 12 months, 18 months and 24 months.
  The change in vit C level from baseline (normal range 4-8.8mg/ L)
Change in fibrosis markers. | Change is assessed baseline, 6 months, 12 months, 18 months and 24 months.
  Change in Nt_ProBNP from the baseline (Normal values up to 381 pg/mL)
Change in inflammation markers. | Change is assessed baseline, 6 months, 12 months, 18 months and 24 months.
  To assess inflammation high sensitivity C reactive protein will be measured by nephelometry. (normal value < 5 mg/L
Change in health-related quality of life | The questionnaire will be applied baseline and every six months up to 24 months.
  This outcome will be measured by the SF 36 questionnaire, themaximun punctuation is 100, as greater punctuation a better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Oliva Mejía-Rodríguez, PhD, Principal Investigator — CIBIMI IMSS
Locations (1):
- Cibimi - Hgz 83 Imss, Morelia, Michoacán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available six months after the end of the study
Access Criteria: Data access request will be reviewed by the research institutional board.